CLINICAL TRIAL: NCT04742803
Title: Face Study of the Effects of Needling Using the Straberi Epistamp for the Improvement of Fine Lines and Skin Laxity.
Brief Title: Straberi Epistamp Needling Treatment For Skin Rejuvenation
Acronym: ESAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universal Skincare Institute (Other)
Collaborators: Lavish Beauty (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1116
Record Dates: First submitted 2020-10-01; First posted 2021-02-08 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Wrinkle; Elastic Skin; Collagen Degeneration
Keywords: microneedling
MeSH Terms: conditions — Ehlers-Danlos Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Straberi Epistamp Needling Treatment (Other): Non-Randomized treatment for patients who seek improvement for elastin, fine lines, deep wrinkles, and collagen production using Straberi Epistamp needling treatment
  Interventions: Device: Straberi Epistamp Microneedling Treatment
- No Treatment (Other): Non-Randomized patients who seek improvement for elastin, fine lines, deep wrinkles, and collagen production.
  Interventions: Device: Straberi Epistamp Microneedling Treatment

INTERVENTIONS:
Device: Straberi Epistamp Microneedling Treatment — The patient's entire face will be treated with the Straberi Epistamp needling device.
  The following settings will be used as a treatment protocol. Needle length between .02- 1.55 mm
  Other Names: Needling

SUMMARY:
This pilot study will expand knowledge and application needling using the Epistamp device for the improvement of a new vitalized epidermal layer with new vibrant active cells, supported by more robust collagen and elastin fine lines, deep wrinkles, and collagen production.

DETAILED DESCRIPTION:
This pilot study will expand the knowledge and application needling using the Epistamp device and its benefits for improving the appearance of fine lines, deep wrinkles, and collagen production. The pilot aims to objectively measure skin quality using the Derma Scan, photographs and provide objective data showing improvement by way of the Universal Skincare Institute Blood Flow Scale.

ELIGIBILITY:
Inclusion Criteria:

* Derma Scan showing aging including skin texture, wrinkles, brown spots, and pores.
* Patients willing to sign informed consent.
* Patients willing to be photographed and video documented
* Patients willing to consent to 3 months of treatment

Exclusion Criteria:

* History of eczema in the treatment area; psoriasis and any other chronic skin conditions
* History of actinic (solar) keratosis in the treatment area;
* History of hemophilia
* History of diabetes
* The presence of raised moles, warts on the targeted area.
* Collagen vascular diseases or cardiac abnormalities
* Blood clotting problems
* Active bacterial or fungal infection
* Facial melanosis
* Malignant tumors
* Immunosuppression
* Use of blood thinners or prednisone
* Corticosteroids within two weeks of the procedure
* Chronic liver disease
* Porphyria or other skin diseases.
* Patient not willing to sign informed consent.
* TCA peels in the last 5 weeks
* Subject currently has moderate to severe acne on the face.
* Microneedling within the last 6 months
* Subject has an active infection.
* Subject has a history of a bleeding disorder
* Subject has a history of keloidal tendency
* Subject has received ablative or non-ablative laser treatments in the previous 6 months.
* Subject has taken Accutane within the previous 3 months.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-23 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-10-12 (Actual)

PRIMARY OUTCOMES:
The Global Aesthetic Improvement Scale (GAIS) | 6 months
  The Global Aesthetic Improvement Scale (GAIS) is a 5-point scale rating global aesthetic improvement in appearance, compared to pretreatment, as judged by the investigator 5 point scale ranging from 1 to 5 with 5 = The appearance has worsen compared with the original condition and 1 = Excellent corrective results investigator.

SECONDARY OUTCOMES:
Overall Skin improvement assessed by Derma Scan | 6 months
  The Derma Scan System utilizes two special lighting systems (RGB +UV) and smart skin analyzer software that allows two images (before and after care) to be compared side by side, which can be used to detect the changes in skin.
Photographs | 6 months
  Digital imaging device using a grid background with controlled lighting and setting to grade acne scar improvement on a quartile grading scale(1 = 1% to 25%, 2 = 26 to 50%, 3 = 51 to 75%, 4 = >76% improvement).
To evaluate the impact on the quality of life (DLQI) | 6 months
  The Dermatology Life Quality Index questionnaire (DLQI) is 10 questions were asked to the patients and score is 0-3 for each question. The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
Wrinkle Severity Rating Scale (WSRS) | 6 months
  The Wrinkle Severity Rating Scale assesses the presence and severity of wrinkles at rest in a rating scale from 0 to 4, where 0 means no visible wrinkles, 1 means minimal wrinkles, 2 means shallow wrinkles, 3 means moderately deep wrinkles and 4 means very deep wrinkles.

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Wright, MD, Principal Investigator — Columbia University/ Harlem Hospital; Leslie L Nesbitt, Study Chair — Universal Skincare
Locations (1):
- Lavish, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Once the overall trial is completed and sensitive detailed information is legally advised to published.

REFERENCES:
- [Background] Goodman GJ, Baron JA. Postacne scarring: a qualitative global scarring grading system. Dermatol Surg. 2006 Dec;32(12):1458-66. doi: 10.1111/j.1524-4725.2006.32354.x. PMID 17199653
- [Background] Finlay AY, Khan GK. Dermatology Life Quality Index (DLQI)--a simple practical measure for routine clinical use. Clin Exp Dermatol. 1994 May;19(3):210-6. doi: 10.1111/j.1365-2230.1994.tb01167.x. PMID 8033378
- See also: Derma Scan — http://universalskincareinstitute.com/